CLINICAL TRIAL: NCT00819117
Title: INvestigation of TRansvenous Versus EPIcarDial Left Ventricular Stimulation Technique
Acronym: INTREPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Angelo Rivetti, Country Manager, St.Jude Medical Italia Spa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR05033IT
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Epicardial leads; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transvenous Lead (TVN CRT) (Active Comparator): Control group: resynchronization via a transvenous left ventricular lead (TVN CRT)
  Interventions: Device: Cardiac Resynchronization Therapy implant
- Epicardial Lead (EPI CRT) (Experimental): Treatment group: resynchronization via an epicardial left ventricular lead (EPI CRT)
  Interventions: Device: Cardiac Resynchronization Therapy implant

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy implant — Device implant with appropriate leads

SUMMARY:
The purpose of this study is to demonstrate that epicardial and transvenous left ventricular leads are safe and effective for cardiac resynchronization therapy in heart failure patients implanted with a CRT device.

DETAILED DESCRIPTION:
This clinical trial is a multicenter, prospective, randomized, parallel, open study designed to compare epicardial left ventricular pacing to transvenous left ventricular pacing for delivering cardiac resynchronization therapy.

After a pre-implant baseline evaluation, patients will be randomized in a 1:1 fashion to one of two groups:

* Control group: resynchronization via a transvenous left ventricular lead (TVN CRT);
* Treatment group: resynchronization via an epicardial left ventricular lead (EPI CRT).

All patients taking part in this study will undergo the implantation of a CRT device with or without ICD back-up (depending on the physician's decision), with right atrial and right ventricular transvenous leads.

Patients will attend protocol scheduled visits before implant (pre-implant baseline evaluation), and post-implant: before hospital discharge, 6 weeks post-implant (optional visit), 3 months (optional visit), and 6 months after implant, time of study termination.

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication for implantation of an CRT device (ESC guidelines , including any update);
* Have a stable pharmacological therapy.

Exclusion Criteria:

* Have a contra-indication to general anesthesia;
* Have a scheduled cardiac surgery;
* Have had a recent myocardial infarction, unstable angina or cardiac revascularization (PTCA or CABG) within 1 month of enrollment;
* Have a life expectancy of less than 6 months;
* Are unable to provide informed consent;
* Are unable to comply with the follow-up schedule and tests;
* Are minor (age below 18 years);
* Are pregnant or are planning for pregnancy in the next 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The efficacy will be evaluated by comparing the pacing thresholds at 6 months between the two groups. The safety will be evaluated by comparing the survival from lead-related complications at 6 months between the two groups. | 6 months follow up after implant

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Bongiorni, MD, Principal Investigator — Ospedale Cisanello, Pisa, Italy
Locations (2):
- Italy (2):
  - Ospedale Cisanello, Pisa
  - Azienda Sanitaria Osperaliera Ordine Mauriziano, Torino